CLINICAL TRIAL: NCT04521153
Title: Camrelizumab Combined With Apatinib Mesylate for Perioperative Treatment of Resectable Hepatocellular Carcinoma：a Randomized, Open-label, Parallel, Multicenter Trial
Brief Title: Camrelizumab Combined With Apatinib Mesylate for Perioperative Treatment of Resectable Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-ZJ-SK-2020
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma; Immunotherapy; Molecular Targeted Therapy
Keywords: Camrelizumab; apatinib mesylate; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Preoperative camrelizumab combined with apatinib mesylate (q2w, 2 cycles) → radical surgery →sequential camrelizumab and apatinib mesylate (q3w, at least 6 cycles). One cycle of postoperative TACE treatment 4-6 weeks after surgery is allowed.
  (Note: Surgery within 2-4 weeks after the last administration of neoadjuvant therapy, postoperative TACE treatment at least 4 weeks after surgery, and camrelizumab combined with apatinib mesylate 4 weeks after surgery or 2-4 weeks after post-operative TACE)
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate; Procedure: Radical surgery
- Control group (Active Comparator): Radical surgery, one cycle of postoperative TACE treatment 4-6 weeks after surgery is allowed.
  (Note: Postoperative TACE treatment at least 4 weeks after surgery)
  Interventions: Procedure: Radical surgery

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab is administered at 200mg, q2w (2cycles) before radical surgery and 200mg, q3w (at least 6 cycles) after radical surgery
  Arms: Experimental group
Drug: Apatinib Mesylate — Apatinib Mesylate is administered at 250mg, qd (2 cycles) before radical surgery and 250mg, qd (at least 6 cycles) after radical surgery
  Arms: Experimental group
Procedure: Radical surgery — Radical surgery

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common primary liver cancer. Hepatectomy is a curable and effective method. However, the recurrence rate is as high as 50%~70% in 5 years after surgery. Perioperative treatment with immunotherapy combined with target therapy is expected to improve the patient's prognosis. This study aims to evaluate the efficacy, safety and tolerability of camrelizumab combined with apatinib mesylate in the perioperative period of resectable hepatocellular carcinoma.The primary purpose of this study is to evaluate the rate of subjects with major pathological response for phase 2 study and event-free survival (EFS) by investigator for phase 3 study of camrelizumab combined with apatinib mesylate in the perioperative period of hepatocellular carcinoma (CNLC Ib-IIIa). The secondary research purpose is to evaluate EFS by Blinded Independent Review Committee, the R0 resection rate, the rate of subjects with major pathological response, the rate of subjects with pathological complete response, overall survival and disease-free survival of camrelizumab combined with apatinib mesylate in the perioperative period of resectable hepatocellular carcinoma. The safety and tolerability is also evaluated.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary liver cancer. Hepatectomy is a curable and effective method. However, the recurrence rate is as high as 50%~70% in 5 years after surgery. Perioperative treatment with immunotherapy combined with target therapy is expected to improve the patient's prognosis. This study aims to evaluate the efficacy, safety and tolerability of camrelizumab combined with apatinib mesylate in the perioperative period of resectable hepatocellular carcinoma. This trial includes subjects with CNLC Ib/IIa/IIb/IIIa HCC. All eligible subjects will be randomized (1:1) to experimental group or control group. In the experimental group, patients will be treated with following: neoadjuvant therapy (camrelizumab and apatinib, 2 cycles), radical surgery, adjuvant therapy (camrelizumab and apatinib, 6 cycles); in the control group, patients will be treated with following: radical surgery. One cycle of postoperative TACE treatment is allowed in both experimental and control group. The primary purpose of this study is to evaluate the rate of subjects with major pathological response for phase 2 study and event-free survival (EFS) by investigator for phase 3 study of camrelizumab combined with apatinib mesylate in the perioperative period of HCC. The secondary research purpose is to evaluate the EFS by Blinded Independent Review Committee, the R0 resection rate, the rate of subjects with major pathological response, the rate of subjects with pathological complete response, overall survival and disease-free survival of camrelizumab combined with apatinib mesylate in the perioperative period of resectable HCC. The safety and tolerability is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this study and sign an informed consent form
2. Age 18~75 years old, no gender limit
3. Hepatocellular carcinoma confirmed by histopathology, cytology or imaging
4. CNLC stage Ib/IIa/IIb/IIIa hepatocellular carcinoma, except for CNLC IIIa hepatocellular carcinoma combined with main portal vein tumor thrombus
5. Child-Pugh score: A grade (≤6 points)
6. ECOG PS score: 0-1 points

Exclusion Criteria:

1. Known intrahepatic cholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and fibrolamellar cell carcinoma; have other active malignancies other than HCC within 5 years or at the same time.
2. Currently accompanied by interstitial pneumonia or interstitial lung disease
3. Existence of active autoimmune disease or history of autoimmune disease and may relapse
4. Patients with active infection, unexplained fever ≥38.5℃ within 1 week before randomization, or baseline white blood cell count >15*10^9/L
5. Patients with congenital or acquired immune deficiencies (such as HIV-infected persons)
6. Those who are known to be allergic to any monoclonal antibodies, anti-angiogenesis targeted drugs or excipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) assessed by investigator | up to 3 years
  The primary endpoint of phase 3 study is EFS assessed by investigator, which is defined as time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, or death due to any cause.
The rate of subjects of major pathological response (MPR) | From enrollment to 30 days post-surgery
  The primary endpoint of phase 2 study is the rate of subjects of MPR in the first 60 patients in the experimental group. MPR is defined as less than or equal to 50% residual tumor after neoadjuvant therapy of camrelizumab and apatinib therapy.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 5 years
  OS is defined as the time from randomisation to death.
EFS assessed by Blinded Independent Review Committee (BIRC) | up to 3 years
  The primary endpoint of phase 3 study is EFS assessed by BIRC, which was retrospectively reviewed by two independent radiologists. EFS is defined as time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, or death due to any cause.
Disease-free survival (DFS) assessed by investigator | up to 3 years
  DFS is defined as the time from randomization until disease recurrence or death from any cause.
R0 resection rate | From enrollment to 30 days post-surgery
  R0 resection rate
The rate of subjects of major pathological response (MPR) | From enrollment to 30 days post-surgery
  The rate of subjects of MPR in all enrolled patients. MPR is defined as less than or equal to 50% residual tumor after neoadjuvant therapy of camrelizumab and apatinib therapy.
The rate of subjects of pathologic complete response (pCR) | From enrollment to 30 days post-surgery
  The rate of subjects of pCR
Safety and tolerability | From enrollment to the end of treatment at 90 days
  The incidence of adverse events, severe adverse events; surgery related safety.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Doctor, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Colombet M, Soerjomataram I, Mathers C, Parkin DM, Pineros M, Znaor A, Bray F. Estimating the global cancer incidence and mortality in 2018: GLOBOCAN sources and methods. Int J Cancer. 2019 Apr 15;144(8):1941-1953. doi: 10.1002/ijc.31937. Epub 2018 Dec 6. PMID 30350310
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Background] Allemani C, Weir HK, Carreira H, Harewood R, Spika D, Wang XS, Bannon F, Ahn JV, Johnson CJ, Bonaventure A, Marcos-Gragera R, Stiller C, Azevedo e Silva G, Chen WQ, Ogunbiyi OJ, Rachet B, Soeberg MJ, You H, Matsuda T, Bielska-Lasota M, Storm H, Tucker TC, Coleman MP; CONCORD Working Group. Global surveillance of cancer survival 1995-2009: analysis of individual data for 25,676,887 patients from 279 population-based registries in 67 countries (CONCORD-2). Lancet. 2015 Mar 14;385(9972):977-1010. doi: 10.1016/S0140-6736(14)62038-9. Epub 2014 Nov 26. PMID 25467588
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Akateh C, Black SM, Conteh L, Miller ED, Noonan A, Elliott E, Pawlik TM, Tsung A, Cloyd JM. Neoadjuvant and adjuvant treatment strategies for hepatocellular carcinoma. World J Gastroenterol. 2019 Jul 28;25(28):3704-3721. doi: 10.3748/wjg.v25.i28.3704. PMID 31391767
- [Background] Takayama T, Sekine T, Makuuchi M, Yamasaki S, Kosuge T, Yamamoto J, Shimada K, Sakamoto M, Hirohashi S, Ohashi Y, Kakizoe T. Adoptive immunotherapy to lower postsurgical recurrence rates of hepatocellular carcinoma: a randomised trial. Lancet. 2000 Sep 2;356(9232):802-7. doi: 10.1016/S0140-6736(00)02654-4. PMID 11022927
- [Background] Lee JH, Lee JH, Lim YS, Yeon JE, Song TJ, Yu SJ, Gwak GY, Kim KM, Kim YJ, Lee JW, Yoon JH. Adjuvant immunotherapy with autologous cytokine-induced killer cells for hepatocellular carcinoma. Gastroenterology. 2015 Jun;148(7):1383-91.e6. doi: 10.1053/j.gastro.2015.02.055. Epub 2015 Mar 4. PMID 25747273
- [Background] Peng BG, Liang LJ, He Q, Kuang M, Lia JM, Lu MD, Huang JF. Tumor vaccine against recurrence of hepatocellular carcinoma. World J Gastroenterol. 2005 Feb 7;11(5):700-4. doi: 10.3748/wjg.v11.i5.700. PMID 15655825
- [Background] Kuang M, Peng BG, Lu MD, Liang LJ, Huang JF, He Q, Hua YP, Totsuka S, Liu SQ, Leong KW, Ohno T. Phase II randomized trial of autologous formalin-fixed tumor vaccine for postsurgical recurrence of hepatocellular carcinoma. Clin Cancer Res. 2004 Mar 1;10(5):1574-9. doi: 10.1158/1078-0432.ccr-03-0071. PMID 15014006
- [Background] Bruix J, Takayama T, Mazzaferro V, Chau GY, Yang J, Kudo M, Cai J, Poon RT, Han KH, Tak WY, Lee HC, Song T, Roayaie S, Bolondi L, Lee KS, Makuuchi M, Souza F, Berre MA, Meinhardt G, Llovet JM; STORM investigators. Adjuvant sorafenib for hepatocellular carcinoma after resection or ablation (STORM): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2015 Oct;16(13):1344-54. doi: 10.1016/S1470-2045(15)00198-9. Epub 2015 Sep 8. PMID 26361969
- [Background] Wang SN, Chuang SC, Lee KT. Efficacy of sorafenib as adjuvant therapy to prevent early recurrence of hepatocellular carcinoma after curative surgery: A pilot study. Hepatol Res. 2014 May;44(5):523-31. doi: 10.1111/hepr.12159. Epub 2013 Jun 13. PMID 23672310
- [Background] Zhang XP, Chai ZT, Gao YZ, Chen ZH, Wang K, Shi J, Guo WX, Zhou TF, Ding J, Cong WM, Xie D, Lau WY, Cheng SQ. Postoperative adjuvant sorafenib improves survival outcomes in hepatocellular carcinoma patients with microvascular invasion after R0 liver resection: a propensity score matching analysis. HPB (Oxford). 2019 Dec;21(12):1687-1696. doi: 10.1016/j.hpb.2019.04.014. Epub 2019 May 29. PMID 31153833
- [Background] Wang D, Jia W, Wang Z, Wen T, Ding W, Xia F, Zhang L, Wu F, Peng T, Liu B, Zhou C, Zheng Q, Miao X, Peng J, Huang Z, Dou K. Retrospective analysis of sorafenib efficacy and safety in Chinese patients with high recurrence rate of post-hepatic carcinectomy. Onco Targets Ther. 2019 Jul 17;12:5779-5791. doi: 10.2147/OTT.S168447. eCollection 2019. PMID 31410023
- [Background] Chen Q, Shu C, Laurence AD, Chen Y, Peng BG, Zhen ZJ, Cai JQ, Ding YT, Li LQ, Zhang YB, Zheng QC, Xu GL, Li B, Zhou WP, Cai SW, Wang XY, Wen H, Peng XY, Zhang XW, Dai CL, Bie P, Xing BC, Fu ZR, Liu LX, Mu Y, Zhang L, Zhang QS, Jiang B, Qian HX, Wang YJ, Liu JF, Qin XH, Li Q, Yin P, Zhang ZW, Chen XP. Effect of Huaier granule on recurrence after curative resection of HCC: a multicentre, randomised clinical trial. Gut. 2018 Nov;67(11):2006-2016. doi: 10.1136/gutjnl-2018-315983. Epub 2018 May 25. PMID 29802174
- [Background] Qin S, Ren Z, Meng Z, Chen Z, Chai X, Xiong J, Bai Y, Yang L, Zhu H, Fang W, Lin X, Chen X, Li E, Wang L, Chen C, Zou J. Camrelizumab in patients with previously treated advanced hepatocellular carcinoma: a multicentre, open-label, parallel-group, randomised, phase 2 trial. Lancet Oncol. 2020 Apr;21(4):571-580. doi: 10.1016/S1470-2045(20)30011-5. Epub 2020 Feb 26. PMID 32112738
- [Background] Xu J, Zhang Y, Jia R, Yue C, Chang L, Liu R, Zhang G, Zhao C, Zhang Y, Chen C, Wang Y, Yi X, Hu Z, Zou J, Wang Q. Anti-PD-1 Antibody SHR-1210 Combined with Apatinib for Advanced Hepatocellular Carcinoma, Gastric, or Esophagogastric Junction Cancer: An Open-label, Dose Escalation and Expansion Study. Clin Cancer Res. 2019 Jan 15;25(2):515-523. doi: 10.1158/1078-0432.CCR-18-2484. Epub 2018 Oct 22. PMID 30348638
- [Derived] Wang Z, Fan J, Zhou S, Sun Y, Liang F, Ji Y, Gu F, Li T, Peng L, Peng T, Huang X, Ding Z, Bai D, Xiang B, Tan G, Wen T, Zeng Y, Han F, Zhang Y, Wu S, Zhao H, Chen Y, Shi G, Hou Z, Sun Y, Zhu W, Zhou J. Perioperative camrelizumab plus rivoceranib versus surgery alone in patients with resectable hepatocellular carcinoma at intermediate or high risk of recurrence (CARES-009): a randomised phase 2/3 trial. Lancet. 2025 Nov 1;406(10515):2089-2099. doi: 10.1016/S0140-6736(25)01720-9. Epub 2025 Oct 19. PMID 41125112